CLINICAL TRIAL: NCT03838146
Title: Influence of Maternal Exercise on Infant Skeletal Muscle and Metabolomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Linda May, Associate Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12-002524b
Record Dates: First submitted 2018-11-05; First posted 2019-02-12 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: comparing 3 exercise interventions to a control (non-exercise) group
Who Masked: Care Provider, Investigator
Masking Description: the clinicians and investigators taking measures are blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-Exercise Control (No Intervention): This group will come in regularly for measurements, but will not have an exercise intervention. If necessary for retention of participants, then we will meet with controls 3 times a week to stress reduction techniques.
- Resistance Type of Exercise (Experimental): This group will participate in resistance exercise intervention 3 times per week from enrollment to delivery.The resistance training (RT) group will perform three sets of 12-15 repetitions of 10-12 resistance exercises in a circuit, with rest of 30-60 seconds between sets as needed. Participants will use a combination of Cybex machines (Cybex International, Medway, MA), resistance bands, and free weights. Routines will change every 3 weeks to add variety and improve compliance.
  Interventions: Behavioral: Types of Exercise
- Combination Type of Exercise (Experimental): This group will participate in combination (aerobic+resistance) exercise intervention 3 times per week from enrollment to delivery. The combination (CT) group will alternate between resistance and aerobic exercises. Participants will perform 4.5 minute bouts of aerobic exercise and perform four resistance exercises of 12-15 repetition that vary between aerobic bouts[17-19]. The aerobic exercise bouts will be performed on the aerobic machine of the participant's choosing as described above. The resistance routine will follow similar guidelines as the resistance group.
  Interventions: Behavioral: Types of Exercise
- Aerobic Type of Exercise (Experimental): This group will participate in aerobic exercise intervention 3 times per week from enrollment to delivery. The aerobic training (AT) group will perform a continuous aerobic exercise of their choosing (e.g., treadmill, ellipticals, stairs, Zumba, or outside walking/jogging). Participants' ability to choose an aerobic activity that they are comfortable with and enjoy is intended to improve compliance.
  Interventions: Behavioral: Types of Exercise

INTERVENTIONS:
Behavioral: Types of Exercise — moderate intensity exercise
  Arms: Aerobic Type of Exercise; Combination Type of Exercise; Resistance Type of Exercise

SUMMARY:
The American Heart Association suggests that heart disease prevention should target pregnancy and the first year of life; however, there is a fundamental gap in knowledge regarding the effects of prenatal exercise on the prevention of heart disease.[1, 2] Insulin resistance in skeletal muscle is believed to be a critical contributor to the metabolic syndrome which increases the risk for cardiovascular disease (CVD). Conversely, exercise improves insulin sensitivity and many other facets of skeletal muscle function and metabolism; however, it is unclear if this positive effect can be "imprinted" in the skeletal muscle of the fetus with maternal exercise and accordingly diminish CVD risk in offspring. Our previous studies found that exercise during pregnancy leads to improved heart measures and reduced adiposity.[3-6] These studies demonstrated the potential for maternal exercise to reduce risk for CVD, but the cellular mechanisms involved, however, are not clearly evident. The proposed project will fill this critical gap and assess the influence of maternal exercise intervention to "imprint" progenitor stem cells in the fetus (umbilical cord tissue) to develop into insulin sensitive skeletal muscle and also improve indices of infant morphometry and movement. Using a randomized design, 160 women will perform either exercise intervention (aerobic training, resistance training, or both) or usual care (controls). Infant cord tissue and blood will be sampled at birth while blood will be sampled at 1 month of age. Similarly, infant neuromotor and morphometric examinations will be performed at 1 month. and at 1-month of age via blood sample, neuromotor, and morphometric examinations. The rationale for the project is to elucidate the effects of maternal exercise on offspring health outcomes and determine specific metabolic targets predictive of offspring long-term disease risk. The investigators will test the central hypothesis that exercise during pregnancy alters skeletal muscle in a manner which decreases the risk of heart disease in offspring. To test this central hypothesis, the investigators will pursue two specific aims: Aim 1- Determine the ability of regular maternal exercise to imprint key myocellular metabolic (insulin sensitivity) properties of offspring mesenchymal stem cells (MSC), neuromotor function, and morphometry. Aim 2- Determine the distinct abilities of regular maternal exercise to imprint the metabolome of offspring MSC.

DETAILED DESCRIPTION:
Is offspring skeletal muscle function and metabolism imprinted by regular maternal exercise? What offspring metabolome markers are altered with regular maternal exercise? The investigators will use a randomized design of 160 women to either exercise intervention (aerobic training, resistance training, or both) or usual care (controls). Infant cord tissue and blood will be sampled at birth while blood will be sampled at 1 month of age. Similarly, infant neuromotor and morphometric examinations will be performed at 1 month. and at 1-month of age via blood sample, neuromotor, and morphometric examinations. The rationale for the project is to elucidate the effects of maternal exercise on offspring health outcomes and determine specific metabolic targets predictive of offspring long-term disease risk.

ELIGIBILITY:
Inclusion Criteria:

* <16 weeks gestation
* singleton pregnancy telephone/email contact

Exclusion Criteria:

* chronic conditions i.e. diabetes, hypertension, HIV, etc.
* use of medications that affect fetal development;
* use of alcohol, tobacco, or other drugs

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — our study focuses on exercise exposure during pregnancy, therefore, all participants are female.
Enrollment: 167 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Human Skeletal Muscles cells grown from MSCs will have insulin responsiveness measured | At Birth
  Western blot analysis of Akt phosphorylation will be conducted on cell lysates from myotubes under basal or following insulin-stimulation. Glycogen synthesis will be measured under basal and insulin-stimulated conditions. Data will be presented as % change in glycogen synthesis following insulin stimulation.

SECONDARY OUTCOMES:
Global and targeted metabolomics analysis will be conducted to map out pathways and mechanisms from regular maternal exercise. Docosahexaenoic acid (DHA), Eicosapentaenoic Acid (EPA), Docosapentaenoic Acid (DPA), and Arachidonic acid (ARA). | At 16 weeks and 36 weeks gestation
  Targeted quantitative LC/MS analysis of DHA and EPA from participants at 16 (pre-training intervention) and 36 weeks, DHA and EPA levels from umbilical cord tissue sample, and DHA and EPA levels from umbilical cord (infant) blood will be compared between groups.
  From our pathway analysis of identified metabolites of interest, we will be able to map the metabolites of interest within common pathways related to maternal exercise exposure.
Peabody Developmental Motor Scales, 2nd edition (PDMS-2) will be performed by a pediatric physical therapist (blinded to group classification) to measure gross motor skills of infants up to 12 months of age. | at 1 month postnatal visit
  3 of the 6 subtests can be used on 1 month olds. All items scored from 0-2, which include:
  1. Reflexes: 8-item subtest that measures child's ability to react to environmental events.
  2. Stationary: 30-item subtest that measures child's ability to control body within center of gravity and retain equilibrium
  3. Locomotion: 89-item subtest that measures child's ability to move from one place to another through crawling, walking, running, hopping, and jumping forward
  we only do the Reflexes Range (0-16), Stationary Range (0-60), and Locomotion Range (0-178) subtests. Each subtest score is also converted to percentile (comparing infant's behavior to the normative sample). All subtest score are summed to determine the Gross Motor Quotient (GMQ), and a GMQ percentile score will be determined.
A trained (blinded) researcher will measure bicep, tricep, and subscapular skinfold measures, circumferences (abdominal, head, mid-upper arm), and lengths (body, femur, leg, humeral). All measures are recorded as mm. | at 1 month postnatal visit
  All measures will be taken in duplicate on the right side following published standards for skinfold and circumference location.
  Data will be used to compare individual skinfolds, sum of skinfolds and circumferences measures between groups
A trained (blinded) researcher will measure body weight on an infant scale | at 1 month postnatal visit
  Body weight will be done to the nearest tenth of a kilogram. Data will be used to compare body weight measures between groups

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
we will not be sharing individual data with other researchers

REFERENCES:
- [Derived] Jevtovic F, Wisseman BL, Jahan F, Claiborne A, Collier DN, DeVente JE, Mouro S, Zeczycki T, Szumilewicz A, Adamo KB, Goodyear LJ, May LE. Maternal exercise alters placental proteome in an exercise mode-specific manner. Am J Physiol Endocrinol Metab. 2025 Dec 1;329(6):E912-E922. doi: 10.1152/ajpendo.00052.2025. Epub 2025 Nov 4. PMID 41187954
- [Derived] Sanchez-Parente S, Kern K, Claiborne A, Wisseman B, Steen D, Roenker B, Lilley A, Strom C, Newton E, DeVente J, Mouro S, Collier D, Kuehn D, Dubose KD, Kelley G, McMillan AG, Castro-Pinero J, Aparicio VA, May LE. Impact of Supervised-concurrent Exercise During Pregnancy on Infant Neuromotor Skills: A Post-hoc Analysis Stratified by Maternal BMI. Sports Med Open. 2025 Jun 20;11(1):78. doi: 10.1186/s40798-025-00886-x. PMID 40542229
- [Derived] Jevtovic F, Claiborne A, DeVente JE, Mouro S, Houmard JA, Broskey NT, May LE. Maternal resistance exercise increases infant energy expenditure. Am J Physiol Endocrinol Metab. 2025 Mar 1;328(3):E354-E361. doi: 10.1152/ajpendo.00414.2024. Epub 2024 Dec 23. PMID 39716848
- [Derived] Jevtovic F, Claiborne A, Biagioni EM, Collier DN, DeVente JE, Mouro S, Kaneko-Tarui T, O-Tierney-Ginn PF, Goodyear LJ, Houmard JA, Broskey NT, May LE. Paternal obesity decreases infant MSC mitochondrial functional capacity. Am J Physiol Endocrinol Metab. 2024 Oct 1;327(4):E441-E448. doi: 10.1152/ajpendo.00239.2024. Epub 2024 Aug 14. PMID 39140975
- [Derived] Jevtovic F, Collier DN, DeVente J, Mouro S, Claiborne A, Wisseman B, Steen D, Kern K, Broskey N, May LE. Maternal exercise increases infant resting energy expenditure: preliminary results. Int J Obes (Lond). 2024 Sep;48(9):1347-1350. doi: 10.1038/s41366-024-01560-0. Epub 2024 Jun 10. PMID 38858465
- [Derived] Jevtovic F, Zheng D, Houmard JA, Kern K, Claiborne A, Lopez CA, Broskey NT, Isler C, DeVente J, Newton E, May LE. Myogenically differentiated mesenchymal stem cell insulin sensitivity is associated with infant adiposity at 1 and 6 months of age. Obesity (Silver Spring). 2023 Sep;31(9):2349-2358. doi: 10.1002/oby.23829. Epub 2023 Aug 8. PMID 37551412
- [Derived] Jevtovic F, Zheng D, Houmard JA, Krassovskaia PM, Lopez CA, Wisseman BL, Steen DM, Broskey NT, Isler C, DeVente J, Fang X, May LE. Effects of Maternal Exercise Modes on Glucose and Lipid Metabolism in Offspring Stem Cells. J Clin Endocrinol Metab. 2023 Jun 16;108(7):e360-e370. doi: 10.1210/clinem/dgad059. PMID 36722208
- [Derived] McDonald SM, Mouro S, Wisseman B, Isler C, DeVente J, Newton E, Hildebrand J, Kuehn D, Kelley G, Chasan-Taber L, Broskey NT, May LE. Influence of prenatal exercise on the relationship between maternal overweight and obesity and select delivery outcomes. Sci Rep. 2022 Oct 15;12(1):17343. doi: 10.1038/s41598-022-22283-0. PMID 36243785